CLINICAL TRIAL: NCT00563095
Title: A Comparative Study of the Efficacy of Transcatheter Arterial Chemoembolization (TACE) and Transcatheter Arterial Pegylated Interferon Embolization (TAIE) for Hepatocellular Carcinoma
Brief Title: A Comparative Study of the Efficacy of Transcatheter Arterial Chemoembolization (TACE) and Transcatheter Arterial Pegylated Interferon Embolization (TAIE) for Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 1942-02; HARECCTR0500039
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Procedure: Transcatheter Arterial Chemoembolization (TACE)
Procedure: Transcatheter Arterial Pegylated Interferon Embolization (TAIE)

SUMMARY:
Primary: To compare the efficacy of TACE and TAIE.

Secondary: To compare the side effects of TACE and TAIE.

The outcome measurements include survival benefit and tumour regression induced by the two therapies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hepatocellular carcinoma not suitable for surgery

Exclusion Criteria:

* Portal vein thrombosis
* Severe arteriovenous shunt
* Bilirubin level > 50 umol/mL
* Prothrombin time > 5 seconds

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-03; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
regression of tumour size | assessment every 6 months

SECONDARY OUTCOMES:
side effects | every treatment given every 8 - 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Man Fung Yuen, Prof, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China